CLINICAL TRIAL: NCT01104584
Title: An Open Label, Multi-center, Phase 3 Study With Corresponding Blinded Image Reading to Determine the Efficacy and Safety of a Single Intravenous Injection of 0.1 mmol/kg Body Weight of Gadobutrol 1.0 Molar (Gadovist®) in Patients With Newly Diagnosed Breast Cancer Referred for Contrast-enhanced Breast MRI
Brief Title: Efficacy and Safety of Gadobutrol 1.0 Molar (Gadovist) for Breast Magnetic Resonance Imaging (MRI)
Acronym: GEMMA 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91782; 2009-009598-90 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Gadobutrol-enhanced MRI; Mammography; Diagnostic Imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadobutrol (Gadavist, BAY86-4875) (Experimental): Patients first received an unenhanced magnetic resonance mammography (MRM), followed by a gadobutrol-enhanced MRM. Gadobutrol was administered at the standard dose of 0.1 mmol/kg body weight (bw) [0.1 ml/kg bw] as an intravenous injection (i.v.) at a rate of 2 ml/sec. Unenhanced MRM (UMRM) and combined unenhanced and contrast (gadobutrol)-enhanced MRM (CMRM) image sets were evaluated in a randomized fashion. After the evaluation of the UMRM or CMRM the respective X-ray mammography (XRM) was added and evaluated together with the UMRM images.
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — A single bolus injection of gadobutrol 1.0 M; 0.1 mmol/kg body weight

SUMMARY:
The purpose of this study is to look at the efficacy (how does it work) and safety of gadobutrol when used for obtaining MR images of both breasts.Women with a recent diagnosis of breast cancer by mammogram (X-ray examination of the breasts) may benefit from MRI of the breasts as MRI may detect additional breast cancers

ELIGIBILITY:
Inclusion Criteria:

* Recent histologically proven diagnosis of breast cancer after having obtained X-Ray Mammography (XRM) of both breasts (according to American College of Radiology [ACR] and performed no longer than 6 weeks prior to enrollment into the study) and has been referred for a contrast-enhanced Magnetic Resonance Mammography (MRM) prior to surgery of the breast.
* if female, a digital XRM is required if any of the following criteria is met:

  * a. patient is younger than 50 years;
  * b. patient has heterogeneously or extremely dense breasts;
  * c. is not post-menopausal (post-menopause defined as at least 12 months prior to inclusion without menstruation).
* if female of childbearing potential, MRM should be performed on the 7-14th day of the menstrual cycle.
* has an estimated glomerular filtration rate (eGFR) value >/= 60 mL/min/1.73m^2 derived from a serum creatinine result within 2 weeks prior to study enrollment.

Exclusion Criteria:

* is a female patient who is pregnant or lactating
* has any contraindication to the MRM examination (e.g. metal implants, phobia) or the use of gadolinium-containing contrast agents.
* has received any contrast agent within 24 hours prior to the study MRM, or is scheduled to receive any contrast agent within 24 hours after the study MRM.
* has severe cardiovascular disease (e.g., known long QT syndrome, acute myocardial infarction [< 14 days], unstable angina, congestive heart failure New York Heart Association class IV) or acute stroke (< 48 hours)).
* has acute renal insufficiency of any severity due to hepato-renal syndrome or in the peri-operative liver transplantation period or who has acute or chronic moderate or severe renal insufficiency (glomerular filtration rate < 60 mL/min/1.73m^2).
* has received chemotherapy or hormonal therapy for breast cancer within 6 months.
* has received hormone replacement therapy within 4 weeks prior to study drug administration.
* is scheduled or likely to require a surgery and/or biopsy in the time period up to 24 hours following study drug application
* has prior excisional biopsy or breast surgery less than 6 months before enrollment and between XRM and study MRM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (42):
- United States (9):
  - Tucson, Arizona
  - Oakland, California
  - Englewood, Colorado
  - Chicago, Illinois
  - New York, New York
  - Columbus, Ohio
  - Providence, Rhode Island
  - San Antonio, Texas
  - Tacoma, Washington
- Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina
- Canada (3):
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (9):
  - Erlangen, Bavaria
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Göttingen, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Bochum, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Gera, Thuringia
  - Berlin
- India (3):
  - Mumbai, Maharashtra
  - Delhi
  - Mumbai
- Netherlands (3):
  - Eindhoven, EJ
  - Maastricht
  - Nijmegen
- Poland (5):
  - Bydgoszcz
  - Gliwice
  - Krakow
  - Szczecin
  - Warsaw
- Spain (5):
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Girona, Girona
  - Alzira, Valencia
  - Córdoba
- Taiwan (4):
  - Taipei, Taiwan
  - Taichung
  - Taipei
  - Taizung

REFERENCES:
- [Derived] Endrikat J, Schmidt G, Haverstock D, Weber O, Trnkova ZJ, Barkhausen J. Sensitivity of Contrast-Enhanced Breast MRI vs X-ray Mammography Based on Cancer Histology, Tumor Grading, Receptor Status, and Molecular Subtype: A Supplemental Analysis of 2 Large Phase III Studies. Breast Cancer (Auckl). 2022 Apr 19;16:11782234221092155. doi: 10.1177/11782234221092155. eCollection 2022. PMID 35462754
- [Derived] Sardanelli F, Newstead GM, Putz B, Jirakova Trnkova Z, Trimboli RM, Abe H, Haverstock D, Rosenberg M. Gadobutrol-Enhanced Magnetic Resonance Imaging of the Breast in the Preoperative Setting: Results of 2 Prospective International Multicenter Phase III Studies. Invest Radiol. 2016 Jul;51(7):454-61. doi: 10.1097/RLI.0000000000000254. PMID 26840494
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 16 May 2010 - 27 Sep 2011
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Participants first received an unenhanced magnetic resonance mammography (MRM), followed by a gadobutrol-enhanced MRM. Gadobutrol was administered at the standard dose of 0.1 mmol/kg body weight (bw) [0.1 ml/kg bw] as an intravenous injection (i.v.) at a rate of 2 ml/sec. Unenhanced MRM (UMRM) and combined unenhanced and contrast (gadobutrol)-enhanced MRM (CMRM) image sets were evaluated in a randomized fashion. After the evaluation of the UMRM or CMRM the respective X-ray mammography (XRM) was added and evaluated together with the UMRM images.
Period: Overall Study
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Started | 460 (screened and enrolled)
Received Treatment | 439 (treatment started)
Fulfilled Requirements of FAS Population | 397
Completed | 437 (study course completed)
Not Completed | 23
Not completed — Study drug never administered | 21
Not completed — Study prematurely discontinued | 2

BASELINE CHARACTERISTICS:
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Participants first received an unenhanced MRM, followed by a gadobutrol-enhanced MRM. Gadobutrol was administered at the standard dose of 0.1 mmol/kg bw [0.1 ml/kg bw] as an i.v. injection at a rate of 2 ml/sec. UMRM and CMRM image sets were evaluated in a randomized fashion. After the evaluation of the UMRM or CMRM the respective XRM was added and evaluated together with the UMRM images.
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 438
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 310
  Asian | 104
  Black | 17
  American Indian/Alaska Native | 1
  Missing | 7
Country [Number; unit: participants]
  Argentina | 19
  Canada | 33
  Germany | 91
  Spain | 66
  India | 63
  Poland | 70
  Taiwan | 36
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Difference of Sensitivity for Detection of Full Extent of Malignant Breast Disease Using CMRM vs UMRM Per Reader
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the clinical investigators and the 3 blinded readers using the respective imaging modality as malignant. Subsequently the sensitivity percentage was calculated based on the mean of the sensitivities across all participants. The difference was calculated as CMRM value minus UMRM value. For ease of expression, the following abbreviations will be used: Magnetic Resonance Mammography (MRM), Unenhanced MRM (UMRM), combined unenhanced and contrast (gadobutrol)-enhanced MRM (CMRM), X-ray mammography (XRM).
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 390 participants in the Full Analysis Set (FAS) who had regions with malignant disease verified by Standard of Truth (SoT).
Measure: Mean (95% Confidence Interval); unit: difference in sensitivity (%)
Arm/Group | CMRM Versus UMRM
Number analyzed (Participants) | 390
difference in sensitivity (%)
  Reader 1 | 15.2 [11.8 to 18.7]
  Reader 2 | 31.9 [27.3 to 36.6]
  Reader 3 | 30.4 [25.8 to 34.9]
  Investigator | 15.9 [12.4 to 19.4]

2. Primary Outcome: Sensitivity for Detection of Full Extent of Malignant Breast Disease Using CMRM vs UMRM Per Reader
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the clinical investigators and the 3 blinded readers using the respective imaging modality as malignant. Subsequently the sensitivity percentage was calculated based on the mean of the sensitivities across all participants.
Time Frame: Immediately before injection and after injection
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: sensitivity (%)
Arm/Group | CMRM | UMRM
Number analyzed (Participants) | 390 | 390
sensitivity (%)
  Reader 1 | 88.6 [86.1 to 91.1] | 73.3 [69.5 to 77.2]
  Reader 2 | 89.0 [86.4 to 91.6] | 57.0 [52.5 to 61.6]
  Reader 3 | 85.5 [82.5 to 88.4] | 55.1 [50.5 to 59.8]
  Investigator | 95.5 [93.9 to 97.1] | 79.5 [75.9 to 83.2]

3. Primary Outcome: Breast Level Specificity of CMRM for Non-malignant Breasts by Reader
Description: A non-malignant breast was defined as false positive (FP), when the reader assessed at least one breast region as malignant. When all breast regions were assessed as non-malignant, the breast was defined as true negative (TN). Breast level specificity was first defined in participant as number of TN-breasts in participant divided by number of non-malignant breasts in participant. Subsequently the specificity percentage was calculated based on the mean of the specificities across all participants who contributed with at least one non-malignant breast.
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 367 participants in FAS; evaluable for specificity were breasts without malignant disease as verified by Standard of Truth (SoT) for which a CMRM assessment was available.
Measure: Mean (95% Confidence Interval); unit: specificity (%)
Arm/Group | CMRM
Number analyzed (Participants) | 367
specificity (%)
  Reader 1 | 91.8 [89.1 to 94.6]
  Reader 2 | 83.9 [80.2 to 87.7]
  Reader 3 | 82.8 [79.0 to 86.7]
  Investigator | 95.4 [93.3 to 97.5]

4. Secondary Outcome: Breast Level Specificity of CMRM Based on Malignant Breasts
Description: A malignant breast was defined as FP, when the reader using the respective imaging modality assessed more breast regions as malignant as were present according to SoT. Otherwise the breast was assessed as TN. Specificity was then defined as TN/(TN+FP).
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 390 participants in FAS; evaluable for specificity were breasts with malignant disease verified by SoT for which an assessment by the imaging modality was available.
Measure: Mean (95% Confidence Interval); unit: specificity (%)
Arm/Group | CMRM
Number analyzed (Participants) | 390
specificity (%)
  Reader 1 | 54.9 [49.9 to 59.8]
  Reader 2 | 47.2 [42.2 to 52.1]
  Reader 3 | 55.5 [50.6 to 60.4]
  Investigator | 93.8 [91.5 to 96.2]

5. Secondary Outcome: Percentage Difference of Participants Whose Index Cancers Were Detected Using CMRM vs UMRM, CMRM vs XRM, and CMRM vs CMRM+XRM
Description: Index cancer was defined as the cancer confirmed by histology prior to inclusion which made the participants eligible for the study. The difference in percentage of participants was calculated as CMRM value minus UMRM value, CMRM value minus XRM value, CMRM value minus CMRM+XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 388 participants in FAS; index cancer was defined as the cancer confirmed by histology prior to inclusion which made the participant eligible for the study.
Measure: Number (95% Confidence Interval); unit: difference in percentage of participants
Arm/Group | CMRM Versus UMRM | CMRM vs XRM | CMRM vs CMRM+XRM
Number analyzed (Participants) | 388 | 388 | 388
difference in percentage of participants
  Reader 1 | 15.5 [11.1 to 19.8] | 19.8 [14.9 to 24.8] | -1.0 [-2.9 to 0.8]
  Reader 2 | 30.2 [25.0 to 35.4] | 13.9 [9.2 to 18.7] | -1.3 [-3.2 to 0.6]
  Reader 3 | 30.9 [25.6 to 36.2] | 12.9 [7.8 to 17.9] | -2.6 [-4.6 to -0.6]
  Investigator | 14.2 [10.4 to 18.0] | 2.3 [-0.0 to 4.6] | -0.5 [-1.8 to 0.9]

6. Secondary Outcome: Percentage Difference of Participants Whose Additional Index Cancers Were Detected Using CMRM vs UMRM, CMRM vs XRM, and CMRM vs CMRM+XRM
Description: Additional cancer was defined as cancer which was present according to SoT, but which was not defined as index cancer, i.e. was not known when the participant was enrolled into the study. The difference in percentage of participants was calculated as CMRM value minus UMRM value, CMRM value minus XRM value, CMRM value minus CMRM+XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: The evaluation was based on the 84 participants in the FAS who had at least one additional cancer region according to SoT.
Measure: Number (95% Confidence Interval); unit: difference in percentage of participants
Arm/Group | CMRM Versus UMRM | CMRM vs XRM | CMRM vs CMRM+XRM
Number analyzed (Participants) | 84 | 84 | 84
difference in percentage of participants
  Reader 1 | 23.8 [12.4 to 35.2] | 42.9 [30.6 to 55.1] | 0.0 [-4.5 to 4.5]
  Reader 2 | 44.0 [31.7 to 56.4] | 48.8 [36.4 to 61.2] | 0.0 [-1.2 to 1.2]
  Reader 3 | 34.5 [22.6 to 46.4] | 26.2 [13.5 to 38.9] | -2.4 [-6.8 to 2.1]
  Investigator | 35.7 [24.3 to 47.2] | 40.5 [28.3 to 52.7] | -1.2 [-4.7 to 2.3]

7. Secondary Outcome: Difference of Confidence in Diagnosis for Breast Region Diagnosis Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM and CMRM+XRM vs XRM by Reader, Participant Level
Description: The investigator and the blinded readers each recorded his/her confidence in diagnosis for each breast region based on a 4-point scale (1 = not confident, 2 = somewhat confident, 3 = confident, and 4 = very confident). For each participant, the mean of the confidence responses for the diagnosed breast regions was calculated, and rounded to the nearest 0.5. The difference was calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference of scores on a scale
Arm/Group | CMRM Versus UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
difference of scores on a scale
  Reader 1 | 0.97 [0.94 to 1.00] | 1.25 [1.19 to 1.31] | -0.23 [-0.28 to -0.19]
  Reader 2 | 0.95 [0.91 to 0.99] | 0.74 [0.69 to 0.79] | 0.04 [-0.01 to 0.09]
  Reader 3 | 1.73 [1.68 to 1.78] | 1.64 [1.57 to 1.70] | 0.67 [0.61 to 0.74]

8. Other Pre Specified Outcome: Sensitivity for Detection of Full Extent of Malignant Breast Disease Using XRM, CMRM+XRM and UMRM+XRM Per Reader
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the reader using the respective imaging modality as malignant. Subsequently the sensitivity percentage was calculated based on the mean of the sensitivities across all participants.
Time Frame: Immediately before injection and after injection
Population: The analyses were performed for a total number of 390 participants who had regions with malignant disease verified by SoT with available assessment by the imaging modality.
Measure: Mean (95% Confidence Interval); unit: sensitivity (%)
Arm/Group | X-ray Mammography (XRM) | CMRM+XRM | UMRM+XRM
Number analyzed (Participants) | 390 | 390 | 390
sensitivity (%)
  Reader 1 | 69.6 [65.8 to 73.4] | 89.6 [87.3 to 92.0] | 82.5 [79.5 to 85.6]
  Reader 2 | 72.9 [69.2 to 76.7] | 90.3 [87.9 to 92.7] | 80.9 [77.6 to 84.1]
  Reader 3 | 73.2 [69.5 to 76.9] | 88.0 [85.3 to 90.6] | 80.1 [76.8 to 83.4]
  Investigator | 89.1 [86.6 to 91.5] | 96.0 [94.6 to 97.5] | 92.1 [90.0 to 94.2]

9. Other Pre Specified Outcome: Breast Level Specificity of in Non-malignant Breasts Using UMRM, XRM, CMRM+XRM and UMRM+XRM by Reader
Description: as for outcome 3
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 367 participants; evaluable for specificity were breasts with no malignant disease verified by SoT for which an assessment of the imaging modality was available.
Measure: Mean (95% Confidence Interval); unit: specificity (%)
Arm/Group | UMRM | X-ray Mammography (XRM) | CMRM+XRM | UMRM+XRM
Number analyzed (Participants) | 367 | 367 | 367 | 367
specificity (%)
  Reader 1 | 94.4 [92.1 to 96.7] | 92.6 [90.0 to 95.3] | 92.2 [89.5 to 94.9] | 94.3 [92.0 to 96.6]
  Reader 2 | 96.6 [94.8 to 98.4] | 90.3 [87.3 to 93.3] | 83.1 [79.3 to 86.9] | 91.0 [88.1 to 93.9]
  Reader 3 | 95.9 [93.9 to 97.9] | 86.1 [82.6 to 89.6] | 83.0 [79.1 to 86.8] | 85.1 [81.5 to 88.8]
  Investigator | 98.1 [96.8 to 98.4] | 97.8 [96.4 to 99.2] | 95.1 [92.9 to 97.2] | 97.5 [96.1 to 99.0]

10. Other Pre Specified Outcome: Breast Level Specificity in Malignant Breasts Using UMRM, XRM, CMRM+XRM and UMRM+XRM by Reader
Description: as for outcome 4
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 390 participants; evaluable for specificity were breasts with malignant disease verified by SoT for which an assessment by the imaging modality was available.
Measure: Mean (95% Confidence Interval); unit: specificity (%)
Arm/Group | UMRM | X-ray Mammography (XRM) | CMRM+XRM | UMRM+XRM
Number analyzed (Participants) | 390 | 390 | 390 | 390
specificity (%)
  Reader 1 | 71.9 [67.5 to 76.4] | 86.8 [83.4 to 90.2] | 52.7 [47.8 to 57.6] | 69.1 [64.5 to 73.7]
  Reader 2 | 76.2 [71.9 to 80.4] | 75.8 [71.5 to 80.0] | 46.5 [41.6 to 51.5] | 65.4 [60.7 to 70.1]
  Reader 3 | 77.6 [73.4 to 81.7] | 69.4 [64.8 to 73.9] | 54.5 [49.6 to 59.4] | 66.9 [62.2 to 71.6]
  Investigator | 96.2 [94.2 to 98.1] | 97.7 [96.2 to 99.2] | 93.8 [91.5 to 96.2] | 96.0 [94.1 to 98.0]

11. Other Pre Specified Outcome: Breast Level Specificity for All Breasts by Imaging Modality and by Reader
Description: A non-malignant breast was defined as FP when the reader assessed at least one breast region as malignant. A malignant breast was defined as FP, when the reader using the respective imaging modality assessed more breast regions as malignant as were present according to SoT. Otherwise the breast was assessed as TN. Specificity was then defined as (N-FP)/N, where N was total number of breasts.
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 395 participants in FAS; evaluable for specificity were breasts with or without malignant disease verified by SoT with available assessments by the imaging modality.
Measure: Mean (95% Confidence Interval); unit: specificity (%)
Arm/Group | UMRM | CMRM | X-ray Mammography (XRM) | UMRM+XRM | CMRM+XRM
Number analyzed (Participants) | 395 | 395 | 395 | 395 | 395
specificity (%)
  Reader 1 | 83.0 [80.6 to 85.5] | 73.0 [70.2 to 75.9] | 89.7 [87.7 to 91.7] | 81.3 [78.8 to 83.8] | 72.0 [69.2 to 74.8]
  Reader 2 | 86.1 [83.7 to 88.4] | 64.9 [61.9 to 68.0] | 83.0 [80.4 to 85.7] | 77.8 [75.1 to 80.6] | 64.3 [61.2 to 67.4]
  Reader 3 | 86.5 [84.1 to 88.8] | 68.6 [65.4 to 71.8] | 77.6 [74.8 to 80.3] | 75.9 [73.0 to 78.9] | 68.1 [64.9 to 71.3]
  Investigator | 96.6 [95.3 to 97.9] | 94.1 [92.4 to 95.8] | 97.1 [95.9 to 98.3] | 96.2 [94.9 to 97.6] | 94.0 [92.2 to 95.7]

12. Other Pre Specified Outcome: Sensitivity Difference in the Determination of Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the reader using the respective imaging modality as malignant. Subsequently the point estimates were calculated based on the mean of the sensitivities across all participants. Regions with malignant disease verified by SoT comprise unifocal and multifocal regions. Difference in sensitivity is calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in sensitivity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 630 | 630 | 630
difference in sensitivity (%)
  Reader 1 | 17.5 [14.2 to 20.8] | 9.5 [1.9 to 17.1] | 24.3 [20.7 to 27.9]
  Reader 2 | 34.9 [30.1 to 39.7] | 12.5 [9.4 to 15.6] | 21.3 [17.6 to 24.9]
  Reader 3 | 32.1 [27.2 to 36.9] | 10.0 [6.9 to 13.1] | 16.5 [13.0 to 20.0]
  Investigator | 19.0 [14.8 to 23.3] | 6.7 [3.7 to 9.6] | 10.5 [5.7 to 15.2]

13. Other Pre Specified Outcome: Sensitivity Difference in the Determination of Unifocal Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the reader using the respective imaging modality as malignant. Subsequently the point estimates were calculated based on the mean of the sensitivities across all participants. The difference in sensitivity is calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in sensitivity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 570 | 570 | 570
difference in sensitivity (%)
  Reader 1 | -5.8 [-11.1 to -0.4] | -12.6 [-17.7 to -7.5] | -10.2 [-15.3 to -5.1]
  Reader 2 | 4.6 [-1.3 to 10.4] | -12.3 [-17.4 to -7.2] | -12.0 [-17.6 to -6.3]
  Reader 3 | 19.5 [14.2 to 24.8] | -1.9 [-6.4 to 2.6] | 6.9 [2.0 to 11.7]
  Investigator | 12.0 [7.7 to 16.2] | 0.2 [-2.8 to 3.1] | 2.3 [-1.4 to 6.0]

14. Other Pre Specified Outcome: Sensitivity Difference in the Determination of Multifocal Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: as for outcome 13
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in sensitivity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 60 | 60 | 60
difference in sensitivity (%)
  Reader 1 | 46.7 [32.7 to 60.6] | 40.0 [26.0 to 54.0] | 65.0 [52.1 to 77.9]
  Reader 2 | 51.7 [37.5 to 65.9] | 35.0 [20.9 to 49.1] | 46.7 [32.2 to 61.1]
  Reader 3 | 31.7 [18.0 to 45.3] | 21.7 [10.3 to 33.1] | 11.7 [-3.5 to 26.8]
  Investigator | 25.4 [14.3 to 36.5] | 21.7 [11.2 to 32.1] | 36.7 [23.2 to 50.1]

15. Other Pre Specified Outcome: Specificity Difference in the Determination of Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: A malignant breast was defined as FP, when the reader using the respective imaging modality assessed more breast regions as malignant as were present according to SoT. Otherwise the breast was assessed as TN. Specificity was then defined as TN/(TN+FP). The difference was calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in specificity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 3197 | 3197 | 3197
difference in specificity (%)
  Reader 1 | -4.1 [-5.3 to -2.9] | -3.9 [-5.1 to -2.8] | -6.7 [-8.0 to -5.4]
  Reader 2 | -8.4 [-9.9 to -7.0] | -5.7 [-7.2 to -4.2] | -7.5 [-9.0 to -6.0]
  Reader 3 | -6.1 [-7.6 to -4.7] | -2.0 [-3.5 to -0.5] | -3.2 [-4.7 to -1.6]
  Investigator | -1.0 [-1.6 to -0.5] | -0.9 [-1.5 to -0.4] | -1.3 [-1.9 to -0.8]

16. Other Pre Specified Outcome: Specificity Difference in the Determination of Unifocal Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: as for outcome 15
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in specificity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 3257 | 3257 | 3257
difference in specificity (%)
  Reader 1 | -3.2 [-4.5 to -1.9] | -3.1 [-4.3 to -1.9] | -5.6 [-7.0 to -4.3]
  Reader 2 | -7.3 [-8.8 to -5.8] | -5.0 [-6.5 to -3.5] | -6.6 [-8.1 to -5.0]
  Reader 3 | -5.4 [-6.9 to -4.0] | -1.6 [-3.1 to -0.1] | -3.1 [-4.7 to -1.6]
  Investigator | -0.4 [-0.9 to 0.1] | -0.4 [-0.9 to 0.1] | -0.5 [-1.1 to 0.1]

17. Other Pre Specified Outcome: Specificity Difference in the Determination of Multifocal Malignant Breast Disease Using CMRM vs UMRM, CMRM+XRM vs UMRM+XRM, and CMRM+XRM vs XRM Verified by SoT, Breast Region Level
Description: as for outcome 15
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in specificity (%)
Units Other Than Participants: breast regions
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (breast regions) | 3767 | 3767 | 3767
difference in specificity (%)
  Reader 1 | -4.4 [-5.7 to -3.0] | -5.3 [-6.5 to -4.0] | -7.5 [-8.8 to -6.1]
  Reader 2 | -6.5 [-8.0 to -5.0] | -6.7 [-8.2 to -5.2] | -8.2 [-9.8 to -6.7]
  Reader 3 | -2.3 [-3.8 to -0.8] | -2.0 [-3.5 to -0.5] | -1.9 [-3.4 to -0.3]
  Investigator | 1.1 [0.3 to 1.9] | -0.7 [-1.4 to 0.0] | -0.7 [-1.5 to 0.1]

18. Other Pre Specified Outcome: Sensitivity of Detection of Multicentric Malignant Disease Verified by SoT, Breast Level
Description: For a single participant the sensitivity was defined as the proportion of malignant breast regions that were recognized by the reader using the respective imaging modality as malignant. Subsequently the point estimates were calculated based on the mean of the sensitivities across all participants. The difference was calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Mean (95% Confidence Interval); unit: difference in sensitivity (%)
Units Other Than Participants: evaluable breasts
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 397 | 397 | 397
Number analyzed (evaluable breasts) | 44 | 44 | 44
difference in sensitivity (%)
  Reader 1 | 47.7 [31.7 to 63.8] | 38.6 [22.9 to 54.3] | 75.0 [62.2 to 87.8]
  Reader 2 | 56.8 [40.9 to 72.8] | 40.9 [23.9 to 58.0] | 61.4 [45.7 to 77.1]
  Reader 3 | 47.7 [31.7 to 63.8] | 31.8 [18.1 to 45.6] | 43.2 [27.2 to 59.1]
  Investigator | 34.1 [18.7 to 49.4] | 31.8 [16.7 to 47.0] | 52.3 [37.5 to 67.0]

19. Other Pre Specified Outcome: Accuracy Difference of Presence of Bilateral Malignant Disease Verified by SoT by Clinical Investigator, Participant Level
Description: The disease state "bilateral malignant disease" was derived from the assessment of the different regions for each breast (right and left) for investigators for each imaging modality (UMRM, CMRM, XRM, UMRM+XRM, and CMRM+XRM) based on the following rule: If the participant had at least one breast with no malignant region , the assessment of bilateral malignant disease was categorized as "No". If the participant had at least one malignant lesion in both breasts, the assessment of bilateral malignant disease was categorized as "Yes". The proportion of correct matches of each different image set to the SoT for the existence of bilateral malignant disease were derived. The analysis was based on the difference in accuracy for the evaluation of bilateral malignant disease for the following image comparisons on a participant level. The difference was calculated as CMRM value minus UMRM value, CMRM+XRM value minus UMRM+XRM value, CMRM+XRM value minus XRM value respectively.
Time Frame: Immediately before injection and after injection
Population: The analyses were based on 380 participants in FAS; evaluable subjects with at least one region verified by SoT in each breast with available CMRM, UMRM, CMRM+XRM, UMRM+XRM and XRM assessment.
Measure: Mean (95% Confidence Interval); unit: difference in accuracy (%)
Arm/Group | CMRM vs UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 380 | 380 | 380
difference in accuracy (%) | 0.5 [-2.0 to 3.1] | -0.3 [-2.5 to 2.0] | -0.8 [-3.2 to 1.6]

20. Other Pre Specified Outcome: Blinded Readers: Inter-reader Agreement on Sensitivity Based on Assessment for UMRM vs CMRM - Breast Region Level
Description: Inter-reader agreement was assessed by considering each breast region to have 2 possibilities (malignant disease / no malignant disease) for an assessment by the 2 image sets (UMRM and CMRM). Kappa value varies from 0 (no agreement) to 1 (perfect agreement).
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Number; unit: Kappa
Units Other Than Participants: breast regions
Arm/Group | CMRM Versus UMRM
Number analyzed (Participants) | 397
Number analyzed (breast regions) | 3827
Kappa | 0.47

21. Other Pre Specified Outcome: Blinded Reader 1: Intra-reader Variability Based on Assessment for CMRM - Breast Level
Description: Intra-reader variability was assessed using a kappa on the match to SoT for the different regions within each participant (match, no match SoT). For each of the 3 readers, intra-reader agreement was assessed by considering each breast region to have 2 possibilities for an assessment by CMRM: matched SoT or did not match SoT. Kappa value varies from 0 (no agreement) to 1 (perfect agreement).
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: Kappa
Units Other Than Participants: evaluable breasts
Arm/Group | CMRM
Number analyzed (Participants) | 397
Number analyzed (evaluable breasts) | 756
Kappa | 0.25

22. Other Pre Specified Outcome: Blinded Reader 2: Intra-reader Variability Based on Assessment for CMRM - Breast Level
Description: as for outcome 21
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: Kappa
Units Other Than Participants: evaluable breasts
Arm/Group | CMRM
Number analyzed (Participants) | 397
Number analyzed (evaluable breasts) | 756
Kappa | 0.23

23. Other Pre Specified Outcome: Blinded Reader 3: Intra-reader Variability Based on Assessment for CMRM - Breast Level
Description: as for outcome 21
Time Frame: Immediately before injection and after injection
Population: All participants in the FAS with assessments for this outcome measure
Measure: Number; unit: Kappa
Units Other Than Participants: evaluable breasts
Arm/Group | CMRM
Number analyzed (Participants) | 397
Number analyzed (evaluable breasts) | 756
Kappa | 0.21

24. Other Pre Specified Outcome: Categorical Accuracy Difference of Extent of Malignant Disease Verified by SoT by Majority Reader, Breast Region Level
Time Frame: Immediately before injection and after injection
Population: The Statistical Analysis Plan (SAP) amendment re-defined study objectives and replaced protocol-defined parameters such as categorical accuracy prior to database closure and breaking the blind. The SAP amendment is based upon review of results of an identical clinical study within the "GEMMA" program and also includes advice from the FDA.
Arm/Group | CMRM Versus UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 0 | 0 | 0

25. Other Pre Specified Outcome: Categorical Accuracy Difference of Extent of Malignant Disease Verified by Histopathology by Majority Reader, Breast Region Level
Time Frame: Immediately before injection and after injection
Population: as for outcome 24
Arm/Group | CMRM Versus UMRM | CMRM+XRM vs UMRM+XRM | CMRM+XRM vs XRM
Number analyzed (Participants) | 0 | 0 | 0

26. Other Pre Specified Outcome: Vital Signs Change From Baseline and Follow-up 24 Hours Post Injection - Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic blood pressure were measured in a supine position. Blood pressure was not to be measured on the arm used for the injection.
Time Frame: Baseline, 24 hours post injection
Population: Safety Analysis Set (SAF): The analysis of safety data was performed using all available data from all participants who administered any amount of gadobutrol.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Patients first received an unenhanced magnetic resonance mammography (MRM), followed by a gadobutrol-enhanced MRM. Gadobutrol was administered at the standard dose of 0.1 mmol/kg body weight (bw) [0.1 ml/kg bw] as an intravenous injection at a rate of 2 ml/sec. Unenhanced MRM (UMRM) and combined unenhanced and contrast (gadobutrol)-enhanced MRM (CMRM) image sets were evaluated in a randomized fashion. After the evaluation of the UMRM or CMRM the respective X-ray mammography (XRM) was added and evaluated together with the UMRM images.
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 432
mmHg
  Systolic blood pressure | -2.7 (15.2)
  Diastolic blood pressure | -2.3 (9.7)

27. Other Pre Specified Outcome: Vital Signs Change From Baseline and Follow-up 24 Hours Post Injection - Heart Rate
Description: Heart rate was measured in a supine position.
Time Frame: Baseline, Follow-up visit (24 hours post injection)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 431
beats/min | -1.7 (10.1)

28. Other Pre Specified Outcome: Number of Participants With at Least One Laboratory Parameter Change From Low or Normal at Baseline to Abnormally High at Follow-up 24 Hours Post Injection
Description: Number of participants with at least one occurrence of changing from low or normal at baseline to high at follow-up.
Time Frame: Baseline, Follow-up visit (24 hours post injection)
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 439
Participants
  Hematology | 41
  Clinical chemistry | 107
  Urinalysis | 144

ADVERSE EVENTS:
Time Frame: Between start of contrast injection and up to 24 hours post-contrast
Description: Treatment-emergent Adverse Events (AEs)
Groups:
- Gadobutrol (Gadavist, BAY86-4875): Participants first received an unenhanced magnetic resonance mammography (MRM), followed by a gadobutrol-enhanced MRM. Gadobutrol was administered at the standard dose of 0.1 mmol/kg body weight (bw) [0.1 ml/kg bw] as an intravenous injection at a rate of 2 ml/sec. unenhanced MRM (UMRM) and combined unenhanced and contrast (gadobutrol)-enhanced MRM (CMRM) image sets were evaluated in a randomized fashion. After the evaluation of the UMRM or CMRM the respective X-ray mammography (XRM) was added and evaluated together with the UMRM images.
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Serious Adverse Events (participants affected / at risk) | 0/439
Other Adverse Events (participants affected / at risk) | 6/439
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=439)
Headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No